CLINICAL TRIAL: NCT00295711
Title: A Multi-Center Double-Blind, Placebo-Controlled Randomized Study of Bicifadine 200 Mg BID, Bicifadine 300 Mg BID, and Bicifadine 400 Mg BID in the Treatment of Chronic Low Back Pain
Brief Title: Efficacy and Safety of Bicifadine in the Treatment of Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DOV Pharmaceutical, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DOV-075-020
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2006-06-23 (Estimated); Status verified 2006-06

CONDITIONS: Chronic Low Back Pain
Keywords: bicifadine; chronic low back pain
MeSH Terms: interventions — bicifadine

INTERVENTIONS:
Drug: Bicifadine

SUMMARY:
The primary objectives of this placebo-controlled clinical trial are to evaluate the analgesic efficacy and safety of bicifadine at three oral dose levels compared with placebo in patients with moderate to severe chronic low back pain.

The secondary objectives are to investigate the dose-response relationship of three dose levels of bicifadine, to evaluate the clinical meaningfulness of bicifadine efficacy, to evaluate the effect of bicifadine on function and general quality of life, to describe the population pharmacokinetics of bicifadine in patients with chronic low back pain, and to evaluate safety following discontinuation of bicifadine treatment.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with low back pain assessed as Class 1, Class 2 or Class 3 according to the Quebec Task Force Classification for Spinal Disorders and without detectable leg weakness on neurological examination.
* Patients must have required on average daily analgesics for the treatment of low back pain for at least 3 months prior to dosing.

Main Exclusion Criteria:

* Patients may not have moderate or severe pain in a location other than the lower back (with the exception of radiation to the lower extremity).
* Patients must not have had lower back surgery within 6 months prior to baseline, nor epidural corticosteroid injections within 3 months prior to baseline.
* Patients may not have an unstable medical condition.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532
Dates: Start 2004-09

PRIMARY OUTCOMES:
- Pain Severity Rating (100 mm visual analog scale)

SECONDARY OUTCOMES:
Short-Form McGill Pain Questionnaire (SF-MPQ)
Roland-Morris Disability Questionnaire (RDQ)
Short-Form 36 (SF-36) Health Survey
Patient's Global Impression of Change (7-point categorical scale)Physician's Global Impression of Change (7-point categorical scale)
Patient's Global Evaluation of Study Medication (5-point categorical scale)
Physician's Global Evaluation of Study Medication (5-point categorical scale)
Incidence of study discontinuation due to lack of efficacy
Plasma PK of bicifadine